CLINICAL TRIAL: NCT04812119
Title: A Neurodevelopmental Data Capture of Patients Diagnosed With CTNNB1 Syndrome With Genotype/Phenotype Gorrelation
Brief Title: Genotype-phenotype Correlations in Children and Adults With CTNNB1 Mutation
Acronym: Gen-Phe CTNNB1
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); National Institute of Chemistry, Ljubljana, Slovenia (Unknown); Children's Medical Research Institute, Westmead, Australia (Unknown); The University of Sydney, Sydney, Australia (Unknown)
Responsible Party: Principal Investigator, Damjan Osredkar, Assoc. Prof. Damjan Osredkar, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-80/2021/3
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: CTNNB1 Gene Mutation
Keywords: CTNNB1 Gene Mutation; CTNNB1 Syndrome; Beta-catenin; Autism Spectrum Disorder; Developmental delay
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with the CTNNB1 mutation: Patient with a diagnosed CTNNB1 mutation.
  Interventions: Diagnostic Test: The Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F); Diagnostic Test: The Autism Spectrum Quotient-Children's Version (AQ-Child); Diagnostic Test: The Autism-Spectrum Quotient (AQ)-Adolescent Version (AQ-Adolescent); Diagnostic Test: The Viking's Speech Scale; Diagnostic Test: The Functional Communication Classification System (FCCS); Diagnostic Test: Brief Infant Sleeping Questionnaire (BISQ); Diagnostic Test: Pediatric Sleep Questionnaire (PSQ); Diagnostic Test: The Eating and Drinking Ability Classification System (EDACS); Diagnostic Test: Mini Manual Ability Classification System (Mini-MACS); Diagnostic Test: Manual Ability Classification System (MACS); Diagnostic Test: The Gross Motor Function Classification System - Expanded and Revised (GMFCS - E&R); Diagnostic Test: The Visual Function Classification System (VFCS); Diagnostic Test: The Early Childhood Oral Health Impact Scale (ECOHIS); Diagnostic Test: The Family Impact Scale (FIS); Diagnostic Test: The Achenbach System of Empirically Based Assessment (ASEBA); Diagnostic Test: Adaptive Behavior Assessment System Third Edition (ABAS-3)

INTERVENTIONS:
Diagnostic Test: The Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F) — The Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F; Robins, Fein, & Barton, 2009) is a 2-stage parent-report screening tool to assess risk for Autism Spectrum Disorder (ASD). It is valid for children 16-30 months old.
  Other Names: M-CHAT-R/F
Diagnostic Test: The Autism Spectrum Quotient-Children's Version (AQ-Child) — The Autism Spectrum Quotient-Children's Version (AQ-Child; Auyeung, Baron-Cohen, Wheelwright & Allison, 2008) is a parent-report questionnaire that aims to quantify autistic traits in children 4-11 years old. It contains 50 likert-type items with responses ranging from "definitely agree" to "definitely disagree".
  Other Names: AQ-Child
Diagnostic Test: The Autism-Spectrum Quotient (AQ)-Adolescent Version (AQ-Adolescent) — The Autism Spectrum Quotient-Children's Version (AQ-Child; Auyeung, Baron-Cohen, Wheelwright & Allison, 2008) is a parent-report questionnaire that aims to quantify autistic traits in children 12-15 years old. It contains 50 likert-type items with responses ranging from "definitely agree" to "definitely disagree".
  Other Names: AQ-Adolescent
Diagnostic Test: The Viking's Speech Scale — The Viking Speech Scale (Pennington, Virella, Mjøen, da Graça Andrada, Murray, Colver, … & Andersen, 2013) is used to classify children's speech production, specifically the ease at which children can make themselves understood using different methods of communication. The scale has four levels and is ordinal. The four levels include: (1) speech is not affected by motor disorder (2) speech is imprecise but usually understandable to unfamiliar listeners (3) speech is unclear and not usually understandable to unfamiliar listeners out of context (3) no understandable speech. It is intended for children above the age of 4 years.
Diagnostic Test: The Functional Communication Classification System (FCCS) — The Functional Communication Classification System (Barty, Caynes & Johnston, 2016) was designed to classify how children with cerebral palsy communicate on a daily basis. The tool focuses on how children typically communicate with familiar and unfamiliar communication partners. There are five classifications a child can be categorized in: (1) effective communicator in most situations (2) effective communicator in most situations, but does need some help (3) an effective communicator in most situations and can communicate small ranges of messages and topics to most familiar people (4) assistance is required in most situations, especially with unfamiliar people and environments. Communicates daily needs and wants to familiar people (5) communicates using undirected movement, vocalisation and/or behaviour, for interpretation by familiar people. The FCCS is valid for use in children up to 13 years.
  Other Names: FCCS
Diagnostic Test: Brief Infant Sleeping Questionnaire (BISQ) — The Brief Infant Sleep Questionnaire (BISQ; Sadeh, 2004) is used to assess sleep patterns, parent perception, and sleep-related behaviors in young children (0-36 months). The BISQ has been validated against actigraphy, daily logs, and has high sensitivity in documenting expected developmental trends in sleep.
  Other Names: BISQ
Diagnostic Test: Pediatric Sleep Questionnaire (PSQ) — Pediatric Sleep Questionnaire (PSQ; Chervin, Hedger, Dillon, Pituch, 2000) has been designed to screen for sleep problems in children. The scale consists of 22 parent-reported items examining snoring and breathing problems, daytime sleepiness, inattention, hyperactivity, and other signs and symptoms of apnea including obesity and nocturnal enuresis. Those questions specifically relate to sleep-disordered breathing (SDB) in children. PSQ has been validated for children 2-18 years old.
  Other Names: PSQ
Diagnostic Test: The Eating and Drinking Ability Classification System (EDACS) — The Eating and Drinking Ability Classification System (EDACS; Sellers, Mandy, Pennington, Hankins, Morris, 2013) has been developed for people with cerebral palsy to describe five distinct levels of ability using the key features of safety and efficiency. The patient can be categorized in: (1) eats and drinks safely and efficiently, (2) eats and drinks safely but with some limitations to efficiency, (3) eats and drinks with some limitations to safety; maybe limitations to efficiency, (4) eats and drinks with significant limitations to safety or (5) unable to eat or drink safely - tube feeding may be considered to provide nutrition. The EDACS is valid for use in children above the age of 36 months.
  Other Names: EDACS
Diagnostic Test: Mini Manual Ability Classification System (Mini-MACS) — The Mini Manual Ability Classification System (Mini-MACS; Eliasson, Krumlinde-Sundholm, 2013) describes how children with cerebral palsy use their hands to handle objects in daily activities. MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life. It has been validated for children 1-4 years of age.
  Other Names: Mini-MACS
Diagnostic Test: Manual Ability Classification System (MACS) — The Manual Ability Classification System (MACS; Eliasson, Krumlinde Sundholm, Rösblad, Beckung, Arner, Öhrvall, Rosenbaum, 2006) describes how children with cerebral palsy use their hands to handle objects in daily activities. MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life. It has been validated for children 4-18 years.
  Other Names: MACS
Diagnostic Test: The Gross Motor Function Classification System - Expanded and Revised (GMFCS - E&R) — The Gross Motor Function Classification System - Expanded & Revised (GMFCS - E&R; Palisano, Rosenbaum, Bartlett, Livingston, 2007) is a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy on the basis of their self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility. Distinctions between levels are based on functional abilities, the need for assistive technology, including hand-held mobility devices (walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement. The questionnaire is available for four age groups of children and youth: 2 to < 4 years, 4 to < 6 years, 6 to < 12 years, and 12 to 18 years.
  Other Names: GMFCS - E&R
Diagnostic Test: The Visual Function Classification System (VFCS) — The Visual Function Classification System (Baranello et al, 2019) is a valid and reliable 5-level classification system of visual functioning for children with Cerebral Palsy. It describes the use of visual abilities in daily life, focusing on activity and participation.
  Other Names: VFCS
Diagnostic Test: The Early Childhood Oral Health Impact Scale (ECOHIS) — The ECOHIS measures the impact of oral problems and/or experience of dental treatment on the quality of life in children under 5 years old and their parents or other family members. It has 13 questions divided into two domains: one related to impact on the child (9 questions), and another to impact on the family (4 questions), measured using the Likert scale. In children with cerebral palsy and/or the ECOHIS has been validated for ages up to 6,5 years, in children with intellectual disability for ages up to 5 years and in children with special need for ages up to 9 years.
  Other Names: ECOHIS
Diagnostic Test: The Family Impact Scale (FIS) — The FIS evaluates the impact of a child's oral condition on family life. It consists of 14 items divided into three subscales: parental/family activity (PA), parental emotions (PE), and family conflict (FC). The financial burden subscale (FB) is the only one that is evaluated separately, since it comprises a single item and addresses economic rather than psychosocial or behavioural impact. It has been validated for children above the age of 12 years.
  Other Names: FIS
Diagnostic Test: The Achenbach System of Empirically Based Assessment (ASEBA) — The Achenbach System of Empirically Based Assessment (ASEBA; Achenbach) is a collection of questionnaires used to assess adaptive and maladaptive behavior and overall functioning in individuals. The system includes report forms for multiple informants - the Child Behavior Checklist (CBCL) is used for caregivers to fill out ratings of their child's behavior, the Youth Self Report Form (YSR) is used for children to rate their own behavior, and the Teacher Report Form (TRF) is used for teachers to rate their pupil's behavior. The ASEBA seeks to capture consistencies or variations in behavior across different situations and with different interaction partners. The ASEBA exists for multiple age groups, including preschool-aged children, school-aged children, adults, and older adults. Scores for individuals in each age group are norm-referenced.
  Other Names: ASEBA
Diagnostic Test: Adaptive Behavior Assessment System Third Edition (ABAS-3) — The ABAS-3 (Harrison, Oakland, 2015) is a rating scale useful for assessing skills of daily living in individuals with developmental delays, autism spectrum disorder, intellectual disability, learning disabilities, neuropsychological disorders, and sensory or physical impairments. Rating forms are filled out by the parent and a teacher. The ABAS-3 covers three broad domains: conceptual, social, and practical, using 11 skill areas within these domains. Tasks focus on everyday activities required to function, meet environmental demands, care for oneself, and interact with others effectively and independently. On a 4-point response scale, raters indicate whether, and how frequently, the individual performs each activity.
  Other Names: ABAS-3

SUMMARY:
The aim of this study is to explore and define the correlations between genotype and phenotype in patients with CTNNB1 mutations as well as monitor and survey the natural history of the CTNNB1 syndrome.

DETAILED DESCRIPTION:
CTNNB1 mutation is linked with autism and other neurodevelopmental disorders. So far, there have been 28 studies published describing 71 patients with this syndrome, which leaves much to be yet discovered. The goal of the study is to reach out to the community and include as many families of patients with CTNNB1 syndrome as possible to create a strong and reliable base of information. the investigators are specifically interested in the correlation between different genotypes and phenotypes and the natural course of the disease. The information gathered with this study will help understand CTNNB1 mutations as well as their effect on patient's overall health and wellbeing. The long-term goal is using this information to help create new treatment options, e.g. gene therapy.

The participants will be guided through a detailed questionnaire about the patient's history, prenatal and delivery risk factors, current medical issues and standardized questionnaires on a variety of subjects that constitute the patient's health and daily function. The investigators wil ask the participants to provide results of genetic testing and other diagnostic measures, thus providing the medical community as well as the families of the patients a reliable overview of the syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosed mutation in the CTNNB1 gene.
* Patients whose parents/caregivers were informed about the aims of the study and have signed the Informed consent form.

Exclusion Criteria:

* Patients who do not have a diagnosed mutation in the CTTNB1 gene.
* Patients whose caregivers have not signed the Informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll and collect data from people who have a diagnosed mutation in the CTNNB1 gene. Participants include people who have a gene change and at least one parent or guardian. Participants can also include multiple people who have a diagnosed CTNNB1 mutation and are within the same family.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Baseline comprehensive collection of medical, behavioral, learning, and developmental information of patients who have documented CTNNB1 gene changes. | Baseline data is collected over the course of one month, on average.
  Patients with a documented CTNNB1 gene change and/or their caretakers will report detailed medical and family history information and provide the results of genetic and other diagnostic testing by completing our online questionnaire. They will be guided through the questionnaire by the help of a medical doctor via an electronic meeting (Zoom) by one of our researchers. Online research surveys will be used to collect information about the patient's genotype and phenotype, with the goal of better understanding the diversity of CTNNB1 syndrome and thus improving clinical care and treatment for these patients.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - The University of Sydney, Sydney
  - Children's Medical Research Institute, Westmead
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No